CLINICAL TRIAL: NCT05498831
Title: Evaluation of a New Pain Management Protocol Involving Intranasal Sufentanil in the Emergency Room : a Prospective Observational Study.
Brief Title: Evaluation of a New Pain Management Protocol Involving Intranasal Sufentanil in the Emergency Room.
Acronym: SUURGE
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Other Study IDs: GHR 1260
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Acute Pain
Keywords: sufentanil; emergencies
MeSH Terms: conditions — Acute Pain; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pain relief protocol according to the recommendations of the French Emergency Medicine Society: The first phase consists in collecting, over a one-month period, data concerning the analgesic management of patients based on the recommendations of the 2010 French Emergency Medicine Society, before the effective implementation of the new pain management protocol, which should be implemented between 2 to 4 months later. Adverse events and patient's satisfaction will also be collected.
  Interventions: Other: Pain assessment at 15 minutes, 30 minutes, 60 minutes, 120 minutes after initial assessment by the triage nurse
- Pain relief protocol with intranasal sufentanil as a starter: The second phase consists in collecting, over a one-month period, data concerning the analgesic management of patients after the implementation of the new protocol based on the use of intranasal sufentanil as a starter for pain of moderate and severe intensity. Adverse events and patient's satisfaction will also be collected during the second phase.
  Interventions: Other: Pain assessment at 15 minutes, 30 minutes, 60 minutes, 120 minutes after initial assessment by the triage nurse

INTERVENTIONS:
Other: Pain assessment at 15 minutes, 30 minutes, 60 minutes, 120 minutes after initial assessment by the triage nurse — Pain will be assessed using a numerical scale

SUMMARY:
Until now, the Mulhouse emergency department used a protocol for severe pain based on morphine titration. In order to relieve patients' pain more quickly, a new protocol was implemented based on the use of intranasal sufentanil.

The primary objective of the study is to prospectively assess the efficacy of the new pain management protocol implemented in the emergency department and based on intranasal sufentanil in combination with paracetamol and codeine for pain of moderate intensity and intranasal sufentanil in combination with paracetamol followed by morphine titration for severe pain. This new pain management protocol has been updated as part of the upcoming French High Authority for Health hospital certification, for which pain management is one of the priority criteria. This research does not change the routine care given to the patient.

DETAILED DESCRIPTION:
Secondary objectives:

1. To assess the rapidity of pain relief with intranasal sufentanil compared to intravenous morphine titration
2. To compare the evolution over time of the pain with the old and new pain management protocol.
3. To assess the safety of sufentanil and morphine titration

Conduct of research:

When a patient is admitted to the Mulhouse emergency department with pain greater than or equal to 4 on the Numerical Scale, the triage nurse or doctor checks the eligibility criteria. If eligible, the nurse or doctor ensures that the patient does not object to the reuse of their data for this research. An information letter is also given to the patient.

Pain will be measured by numerical rating scale at initial assessment by the triage nurse (baseline), at 15mins, 30mins, 60mins and 2hours.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to the Emergency Department of Mulhouse with a numerical pain rating scale > 3 ;
* Patient who did not receive any analgesic except paracetamol in the 4 hours prior to admission ;
* Initial pain assessment with the triage nurse ;
* Patient does not object to the collection of data for the study.

Exclusion Criteria:

* Patient admitted directly to the shock room ;
* Initial pain assessment not performed in triage zone ;
* Numerical Scale > 3 not corroborated by caregiver assessment: Algoplus <2
* Onset of pain after triage nurse visit ;
* Patient with drug intoxication, altered consciousness, alcohol or drug use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Mulhouse emergency department with pain greater than or equal to 4 on the Numerical Scale
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with effective pain relief 30 minutes after initial assessment by nurse | 30 minutes
  Pain relief will be defined as numeric pain rating scale ≤ 3

SECONDARY OUTCOMES:
Time from initial pain assessment by nurse to administration of intranasal sufentanil compared to Intravenous morphine titration | 2 hours
Number of adverse events | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Rottner, MD, Principal Investigator — Groupe Hospitalier de la Région de Mulhouse et Sud-Alsace
Locations (1):
- Hôpital Emile Muller (GHRMSA), Mulhouse, France

IPD SHARING:
Plan to Share IPD: No